CLINICAL TRIAL: NCT07154056
Title: Prospective, Longitudinal, Single-arm Interventional Study Evaluating the Efficacy of Spinal Transforaminal NeuroStimulation (STNS) With FAST and MULTIWAVE Stimulation in Patients With Refractory Chronic Neuropathic Pain
Brief Title: Evaluation of the Efficacy of STNS With FAST and MULTIWAVE in Patients With Refractory Chronic Neuropathic Pain
Acronym: FORASTIM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-A00462-47
Record Dates: First submitted 2025-07-16; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Chronic Neuropathic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lead(s) implantation, 7days trial phase, Implantable Pulse Generator implantation (Experimental): One or two 8-contact lead(s) will be radiologically positioned within the spinal foramen under awake anesthesia in order to optimize paresthesia coverage. This will be followed by a trial phase for a period of 7 days in order to assess the benefits of stimulation. Patients who succeeded the trial phase (at least 30% reduction of leg pain measured with a 5-day pain diary) will be implanted with a permanent system (Implantable Pulse Generator).
  At first, all patients will be programmed under FAST stimulation for at least 24h to fully perceive its efficacy. If the patient is satisfied with FAST then the patient will continue with this program but if the patient is not satisfied, then the patient could switch to other waveforms that will be pre-programmed during the visit including conventional and microburst stimulation.
  Interventions: Device: Lead(s) and Implantable Pulse Generator implantation

INTERVENTIONS:
Device: Lead(s) and Implantable Pulse Generator implantation — 8-contact lead(s) will be radiologically positioned within the spinal foramen under awake anesthesia in order to optimize paresthesia coverage. Awake anesthesia will allow patients to be tested during the surgery in order to determine the sweet spot and the optimal paresthesia coverage using the PREDI-P platform for a single lead. A trial phase will be performed for a period of 7 days in order to assess the benefits of stimulation according to the HAS (French Health Authority) guidelines. Subjects who succeed the lead trial will receive a permanent implant depending on the patient electrical consumption during the lead trial period or according to the implanter decision.

SUMMARY:
The goal of the study is to demonstrate Spinal Transforaminal NeuroStimulation effectiveness with FAST and other waveforms / combinations to relief neuropathic peripheral pain in chronic neuropathic pain patients, at low risk and low energy consumption.

ELIGIBILITY:
Inclusion Criteria:

* Subject has ≥ 18 years and ≤ 80 years
* Subject has a global Visual Analogic Scale ≥ 5
* Subject has non-cancer pain with a significant neuropathic component for at least 6 months.
* Subject has stable pain for at least 30 days
* Pain medication(s) dosage(s) is/are stable for at least 30 days
* Subject is eligible for Spinal Transforaminal NeuroStimulation after a pre-implantation assessment by a multidisciplinary team, as described by the French National Authority for Health (Haute Autorité de Santé)
* Subject understands and accepts the constraints of the study and is able to use the equipment.
* Patient is covered by French national health insurance.
* Subject has given written consent to the study after having received clear and complete information.

Non-inclusion Criteria:

* Subject has a coagulation disorder
* Subject is or has been treated with SCS, subcutaneous or peripheral nerve stimulation, an intrathecal drug delivery system
* Subject has had corticosteroid therapy within the past 30 days
* Subject has had radiofrequency therapy within the past 3 months
* Subject has been diagnosed with cancer in the past 2 years
* Subject has had a spinal surgery within the past 6 months
* Simultaneous participation to any interventional study on health product or any study able to interfere with the current study endpoints.
* Subject has at least one of brain MRI contraindications such as : intracranial clips /Vascular clips/Pace maker/Heart battery, Defibrillator, Implanted Holter (REVEAL type), Neuro-stimulator not compatible with 1.5 T MRI/Stents/ Coils/Cardiac valves (heart)/ Shunt valve/Implanted injection pump/Cochlear implants/Implantable chamber (PAC)/Intracorporeal metal shards/ metallic foreign bodies, the location and the presence of implanted neurostimulation components that are not listed as MRI Conditional, cardiac implantable electronic device, metallic intraocular foreign bodies, cochlear implants, drug infusion pumps, catheters with metallic components, cerebral artery aneurysm clips, magnetic dental implants, tissue expander, artificial limb, hearing aid, piercing.
* Subjects requiring closer protection, i.e. minors, subjects deprived of their freedom by a court or administrative decision, subjects admitted to a health or social welfare establishment, major subjects under legal protection, and finally patients in an emergency setting
* Pregnant or breastfeeding women, women at age to procreate and not using effective contraception.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome for evaluating pain-related health is the mean absolute change in Multidimensional Clinical Response Index. | 6 months
  The Multidimensional Clinical Response Indexwas previously developed and validated to evaluate the pain-related health state of PSPS-T2 patients. This weighted composite outcome includes pain intensity, functional disability, quality of life, psychological distress and pain mapping surface.
  The Multidimensional Clinical Response Indexis a score that ranges from 0 (worst pain-related health status) to 10 (best pain-related health status). The score has been used in several studies evaluating efficacy of different neurostimulation modalities.

SECONDARY OUTCOMES:
Absolute change in pain intensity between baseline and 1-, 3- and 6-month post-Spinal Transforaminal NeuroStimulation follow-up. | 6 months
  Will be used : Pain Visual Analogic Scale (VAS). Pain intensity is measured on a 0-10 scale (0 = no pain ; 10 = worst possible pain).
Evaluation of patient satisfaction at 1-, 3- and 6-month post-Spinal Transforaminal NeuroStimulation. | 6 months
  Patient satisfaction will be assessed using patient Global Impression of Change questionnaire (PGIC).
To evaluate the effects of Spinal Transforaminal NeuroStimulation on neuropathic pain symptoms. | 6 months
  Evaluation of intensity of each symptom (numbness, burning sensation, tingling, allodynia, electric shock, hypoesthesia) using the PainDetect questionnaire.
Surface (cm²) of each symptom calculated using the Pain mapping software. | 6 months
  To evaluate the effects of Spinal Transforaminal NeuroStimulation on neuropathic pain symptoms.
To characterize the Spinal Transforaminal NeuroStimulation neural targeting based on 3D-imaging and electrophysiological exploration in order to precisely identify the optimal paresthesia-based neural target locations. | 6 months
  Imaging data (3D-MRI and CT fusion) pre-operatively to identify the ganglion position related to the foramen at baseline. For electrophysiological data, we will collect lead performance and selectivity for each program used by the patient under paresthesia-based stimulation at 1-, 3- and 6-month follow-ups.
Rate of serious and non-serious adverse events and device deficiencies will be reported. | 6 months
Rate of patients undergoing FAST stimulation (exclusively or in combination with other waveforms) at 6-month follow-up. | 6 months
Mean absolute change in Multidimensional Clinical Response Index for the subgroup of patients undergoing FAST at 1-, 3- and 6-month follow-ups. | 6 months
Absolute change in pain surface between baseline and 1-, 3- and 6-month post-Spinal Transforaminal NeuroStimulation follow-up. | 6 months
  Pain surface will be assessed using the surface of the painful zone (cm²) measured using the pain mapping software.
Absolute change in health related quality of life between baseline and 1-, 3- and 6-month post-Spinal Transforaminal NeuroStimulation follow-up. | 6 months
  Health related quality of life will be assessed using EuroQuol 5 Dimensions 5 levels (EQ5D 5L) index (-0.53 to 1 score ; 1 = full health and 0 = a state as bad as being dead).
Absolute change in functional disability between baseline and 1-, 3- and 6-month post-Spinal Transforaminal NeuroStimulation follow-up. | 6 months
  Functional disability will be assessed using the Oswestry Disability Index (ODI) (0 to 100 score with 0-20 = minimal disability, 21-40 = moderate disability, 41-60 = severe disability, 61-80 = cripple, pain impinges on all aspects of patient's life, 81-100 = patients are bed-bound or exaggerating their symptoms).
Absolute change in anxiety and depression between baseline and 1-, 3- and 6-month post-Spinal Transforaminal NeuroStimulation follow-up. | 6 months
  Anxiety and depression will be assessed using the Hospital Anxiety and Depression Scale (HADS) anxiety and depression scores.
Evaluation of energy consumption at 1-, 3- and 6-month post-Spinal Transforaminal NeuroStimulation. | 6 months
  Energy consumption will be calculated as the delivered electric current (µC per second).

CONTACTS AND LOCATIONS:
Locations (1):
- Poitiers University Hospital, Poitiers, France